CLINICAL TRIAL: NCT05680831
Title: Pulmonary and Inflammatory Responses Following Exposure to a Low Concentration of Ozone or Clean Air for 6.6 Hours With Moderate Exercise in Healthy Young Adults
Brief Title: Pulmonary and Inflammatory Responses Following Exposure to a Low Concentration of Ozone or Clean Air
Acronym: LOCONOZ2
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Martin W. Case (U.S. Federal Agency)
Collaborators: University of North Carolina (Other)
Responsible Party: Sponsor-Investigator, Martin W. Case, Clinical Studies Coordinator, Environmental Protection Agency (EPA)
Organization: Environmental Protection Agency (EPA) (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB# 21-3193
Record Dates: First submitted 2022-12-16; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Lung Injury, Acute; Symptoms and Signs; Neutrophilia Acute
Keywords: lungs; ozone concentration; exercise; inflammation; symptoms
MeSH Terms: conditions — Acute Lung Injury; Signs and Symptoms; Motor Activity; Inflammation

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, cross-over study with two arms.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: TRC Environmental Corporation, who is on-site contractor responsible for the exposure operation will randomize the subjects into either air or ozone arms, neither subjects nor staff involved in conduct of experiments will be informed of exposure conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 0.070 ppm ozone concentration (Experimental): Exposure to 0.070 ppm ozone for 6.6 hours while performing moderate intermittent exercise.
  Interventions: Biological: 0.070 ppm ozone concentration
- Clean air (0.0 ppm ozone) (Experimental): Exposure to clean air (0.0 ppm ozone) for 6.6 hours while performing moderate intermittent exercise.
  Interventions: Biological: Clean air (0.0 ppm ozone)

INTERVENTIONS:
Biological: 0.070 ppm ozone concentration — The concentration of ozone a subject will randomly receive on a visit for 6.6 hours in a controlled atmospheric chamber while performing moderate intermittent exercise.
  Arms: 0.070 ppm ozone concentration
Biological: Clean air (0.0 ppm ozone) — Same subject will randomly receive clean air on another visit separated by at least one week for 6.6 hours in the same controlled atmospheric chamber while performing moderate intermittent exercise.
  Arms: Clean air (0.0 ppm ozone)

SUMMARY:
Purpose: The primary purpose of this study is to measure pulmonary function, symptoms, and pulmonary inflammatory responses in healthy young adults during and immediately after exposure to a low concentration of ozone (0.070 ppm) or clean air for 6.6 hours while undergoing moderate intermittent exercise. This concentration is the current EPA NAAQS standard for ozone.

DETAILED DESCRIPTION:
Potential health effects of ozone have been extensively studied over decades at various levels of exposure concentration and for varying time periods in young healthy adult subjects. Effects of ozone have been well documented particularly for decrements of lung function and an influx of neutrophils and other markers of pulmonary inflammation. The majority of those studies were done at ozone concentrations between 0.12 and 0.40 ppm, considerably higher than the current EPA NAAQS ozone standard of 0.070 ppm, and at exposure durations of two hours, even though the current standard is an 8-hour standard. However, a small number of studies have assessed changes in lung function following exposure to low levels of ozone for several hours. These latter studies have shown that exposure to ozone for 6.6 hours at concentrations between 0.06 and 0.08 ppm causes mild reversible decrements in lung function (1.7-10%) as measured by forced vital capacity (FVC) and forced expired volume at 1 s (FEV1) immediately after exposure in healthy young adults. In addition, in one study an increase in ozone-induced neutrophils was seen in induced sputum following exposure to 0.06 ppm ozone (8) and in bronchoalveolar lavage fluid) following exposure to 0.08 ppm ozone (9). The EPA is considering whether the current ozone NAAQS standard at 0.070 is protective and has asked EPA researchers to conduct a study similar to those done at 0.06 and 0.08 ppm.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women between 18 and 35 years of age.
2. Physical conditions allowing sustained moderate exercise for 6.6 hours.
3. Normal lung function (NHANES III):

   1. FVC > 80 % of that predicted for gender, ethnicity, age and height.
   2. FEV1 > 80 % of that predicted for gender, ethnicity, age and height.
   3. FEV1/FVC ratio > 80 % of predicted values
4. Oxygen saturation > 94 %.
5. Total symptom Score no greater than 20 (out of a possible 60-see accompanying score sheet) with a value no greater than 3 for any one score. No more than one score may be equal to 3.

Exclusion Criteria:

1. Individuals with a diagnosis of COVID-19 and/or hospitalized for COVID-19.
2. Individuals who are not "up to date," [meaning a person has received all recommended COVID-19 vaccines, including any booster dose(s) when eligible with their COVID vaccines as defined by the CDC.]
3. A history of acute and chronic cardiovascular disease, chronic respiratory disease, diabetes,rheumatologic diseases, immunodeficiency state.
4. An acute respiratory illness within 4 weeks.
5. Subjects who are asthmatic or have a history of asthma.
6. Allergic to chemical vapors or gases.
7. Any allergic symptoms during the time of participation in the study
8. Female subjects who are currently pregnant, attempting to become pregnant or breastfeeding
9. Subjects currently taking mega doses of vitamins and supplements, homeopathic/naturopathic medicines or medications which may impact the results of the ozone challenge or interfere with any other medications potentially used in the study (to include systemic steroids and beta blockers). Medications not specifically mentioned here may be reviewed by the investigators prior to a subject's inclusion in the study.
10. Current and past smokers within 2 years, or subjects with a smoking history of at least a pack of cigarettes a day for more than 10 years over your lifetime. This includes vaping, hookah,and e-cigarettes.
11. Uncontrolled hypertension (> 140 systolic, > 90 diastolic). Blood pressure readings equal to or greater that 140 Systolic and equal to or greater that 90 diastolic.
12. Subjects who do not understand or speak English
13. Unspecified illnesses, which in the judgment of the investigator might increase the risk associated with ozone inhalation challenge or exercise, will be a basis for exclusion.

Temporary exclusion criteria:

1. Individuals who have had an acute respiratory illness within 4 weeks.
2. Individuals who have active allergies.
3. Individuals that have engaged in strenuous exercise within 24 hours of any study visit.
4. Individuals unable to avoid drinking alcohol for 24 hours prior to all study visits.
5. Individuals who have been exposed to smoke and fumes for 24 hours before all visits.
6. Individuals that have used an ozone-based home air purifier for 24 hours before all visits.
7. Individuals that have eaten or drank anything for 2 hours prior to the sputum training/screening day visit.
8. Individuals should avoid caffeine for 12 hours prior to all study visits.
9. Individuals should refrain from all over the counter anti-inflammatory agents including those for allergies, and anti-inflammatory drugs or antioxidants for a period of one week prior to the train and to the exposure.
10. Individuals that have been exposed to or have consumed any agent or have undertaken any activity within 24 hours of any study visit that the investigators believe may compromise the results of the study.

    -

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
FVC | measured (pre) before starting 6.6 hours of exercise
  forced vital capacity
Change in FVC | change measured (post) immediately after 6.6 hours of exercise
  change in forced vital capacity
FEV1 | measured (pre) before starting 6.6 hours of exercise
  forced expiratory volume in 1 second
Change in FEV1 | change measured (post) immediately after 6.6 hours of exercise
  change in forced expiratory volume in 1 second

SECONDARY OUTCOMES:
% neutrophils collected by induced sputum | baseline: training/qualification day
  Subjects will breathe a hypertonic saline solution from an ultrasonic nebulizer through a mouthpiece at saline concentrations of 3%, 4%, and 5%. After each inhalation period subjects be asked to cough up the expectorate in a sterile cup for analysis of neutrophil cells influx
change in % neutrophils collected by induced sputum | 18 hours post exposure
  Subjects will breathe a hypertonic saline solution from an ultrasonic nebulizer through a mouthpiece at saline concentrations of 3%, 4%, and 5%. After each inhalation period subjects be asked to cough up the expectorate in a sterile cup for analysis/quantitation of neutrophil cells influx

CONTACTS AND LOCATIONS:
Overall Officials: Andy Ghio, M.D., Principal Investigator — EPA/ORD/CPHEA/PHITD/CRB
Locations (1):
- EPA Human Studies Facility, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No